CLINICAL TRIAL: NCT06704997
Title: Machine Learning Predictive Analysis of Key Factors Influencing Rehabilitation Length of Stay (RLOS) and Direct Hospitalization Costs for Neurological Inpatient Rehabilitation at Tertiary Care Hospital
Brief Title: Machine Learning to Predict Factors Affecting Rehabilitation Length of Stay and Healthcare Costs for Neurological Rehabilitation
Status: Active, not recruiting | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Chua Sui Geok, Karen, Senior Consultant Dr ( MD), Tan Tock Seng Hospital
Other Study IDs: DSRB 2023/00873
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Acquired Brain Injury; Traumatic Brain Injury; Brain Tumor; Central Nervous System Infections; Polytrauma
Keywords: Rehabilitation; Length of Stay; Stroke; Traumatic Brain Injury; Brain tumour; Cancer; Trauma; Acquired Brain Injury; Healthcare; Hospitalisation costs
MeSH Terms: conditions — Stroke; Brain Injuries; Brain Injuries, Traumatic; Brain Neoplasms; Central Nervous System Infections; Multiple Trauma; Neoplasms; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with tertiary neurological rehabilitation: Patients with confirmed diagnosis of stroke, acquired brain injuries, traumatic brain injuries, brain tumours, central nervous system infections and polytrauma from acute neurological or neurosurgical units in Singapore. The cohort will be selected from the TTSH Rehabilitation Centre (TTSH RC) admissions from year 2016 to the present.

SUMMARY:
The aim of this retrospective study is to ascertain total direct costs, rehabilitation length of stay (RLOS) and factors associated with RLOS for neurological inpatient rehabilitation at the tertiary care hospital.

DETAILED DESCRIPTION:
The aim of the study is to identify factors that influence RLOS and the correlated costs for neurological rehabilitation in tertiary rehab using data extracted from EPIC. It is also aimed to identify the median direct costs to find out the main contributors to the costs in the local population. Lastly, the study aims to utilise artificial intelligence or machine learning to analyse the compiled data to develop a predictive model. The model aspires to understand factors associated with extended RLOS and to predict RLOS of patients who require neurological rehabilitation, aiding preemptive measures.

ELIGIBILITY:
Inclusion Criteria:

• All patients who completed inpatient rehabilitation with the index conditions in their discharge summaries

Exclusion Criteria:

• Did not complete inpatient rehabilitation as they are discharged against medical advice

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have admitted to the rehabilitation ward during their inpatient episode for neurological rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rehabilitation length of stay | 1998-2022
  Duration of which patient is admitted to and discharge from the rehabilitation ward.
Hospital bill | 2012-2022
  Bill size of patient's stay in the rehabilitation ward, including subsidies, insurance and copayment.
Housing type | 2014-2023
  Type of housing to look at the socio-economics status of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Karen Chua, MBBS, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
PI need to verify the quality of the data as extraction will involve accessing Ministry of Health government website to obtain deidentified data set